CLINICAL TRIAL: NCT04788212
Title: Adaptation of a Transdiagnostic Behavioral Activation Telehealth Group for Autistic Adults
Brief Title: Transdiagnostic Group Behavioral Activation for Autistic Adults
Acronym: GBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Vanessa H. Bal, PhD, Karmazin & Lillard Chair in Adult Autism; Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020001634
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Autism Spectrum Disorder; Depression, Anxiety; Anxiety; Anger
MeSH Terms: conditions — Autism Spectrum Disorder; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 8 participants with autism and depression, anxiety or anger will participate
Masking Description: This is an open trial feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GBAT (Experimental): 10-week behavioral activation treatment group.
  Interventions: Behavioral: Group Behavioral Activation Therapy for Autism Spectrum Disorder

INTERVENTIONS:
Behavioral: Group Behavioral Activation Therapy for Autism Spectrum Disorder — This will be a modification of the Group Behavioral Activation Therapy program (Chu et al., 2009) for treatment of depression, anxiety and/or anger in autistic adults.

SUMMARY:
The purpose of this study is to evaluate the feasibility, acceptability and effectiveness of a telehealth Group Behavioral Activation Therapy (GBAT) for autistic adults.

DETAILED DESCRIPTION:
Detailed Description: This study is being done to demonstrate the feasibility, acceptability and effectiveness of a telehealth Group Behavioral Activation Therapy (GBAT) for autistic adults. GBAT is intended to help adults manage stress, anxiety, down moods, and anger. Similar programs have been shown to be effective in other contexts but has not yet been used for autistic adults or delivered via telehealth. Because this is a new intervention, the investigators are interested in learning 1) whether GBAT can be done with autistic adults (feasibility), 2) what autistic adults think about GBAT (acceptability), and 3) whether GBAT is effective for helping autistic adults cope with their feelings. Results from this study will be used to inform adaptation to the intervention and planning for future studies to further explore its effectiveness. For this initial feasibility study, 8 autistic adults (18-40 years old) with VIQ and NVIQ>85, reading composite at least 6th grade level and elevated symptoms of depression, anxiety or anger will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18-40 years old
2. Have a confirmed diagnosis of Autism Spectrum Disorders (ASD).
3. Have access to a device (e.g., computer with a webcam or smartphone) in order to complete online surveys and participate in the telehealth videoconferencing sessions
4. *Have a VIQ and NVIQ of 85 or above
5. *Have at least a 6th grade reading composite
6. *Have elevated symptoms of depression, anxiety or anger. This will be determined based on scoring above the borderline or mild threshold on at least one of 3 screening measures (MINI; ASR; DASS-21).

Exclusion Criteria:

1. Are younger than 18 years old, or older than 40 years old (Children are excluded because the focus is on adapting GBAT for adults; Individuals above 40 are excluded to restrict the adult focus to young adults that are more likely to be in similar life stages).
2. Do not have an ASD diagnosis (because the study as the purpose of the current research is to examine GBAT's feasibility with autistic adults).
3. Both VIQ and NVIQ below 85 OR less than 6th grade reading level
4. Do not have elevated scores of depression, anxiety, or anger on the symptom screening measures.
5. Are unable to understand English fluently (because the instruments being investigated are currently only validated in English and the intervention will be delivered in English).
6. Are currently enrolled in another behavioral therapy or psychotherapy targeting depression,
7. the PI's clinical judgment that it would not be in the adult's best interest to be enrolled (e.g., due to factors that may affect their engagement or comfort in the group).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Change in symptoms on the Adult Self Report (ASR) | 10 week study period; 4 week post-treatment
  The ASR is a an assessment of adult psychopathology (e.g., anxiety, depression symptoms). Most of the items are on a 3 point scale including: (0) Not true, (1) Somewhat or sometimes true, and (2) Very often or often true.
Change in Clinician Global Impairment rating | 10 week study period;
  The CGI is a 7 point scale on which the clinician rates the severity of the client's impairment. The scale ranges from 1 (Normal, not at all ill) to 7 Extremely Ill; higher scores indicate more impairment.

SECONDARY OUTCOMES:
Change in symptoms on the Depression Anxiety Stress Scales-21 | 10 week study period; 4 week post-treatment
  The DASS-21 is a 21-item measure of depression and anxiety symptoms. The measure produces scores in 3 domains: depression, anxiety, and stress. The score ranges on each domain is from 0-42. Higher scores on each domain indicate more impairment/ severity.
Change in distress on Patient Health Questionnaire (PHQ-9) | 10 week study period
  The PHQ-9, assessed weekly, is a 9-item questionnaire of psychological function over the past week with all items on a "0" (not at all) to "3" (nearly every day) scale. Total scores range from 0 to 27; higher scores reflect greater levels of depressive symptoms.
Change in anxiety symptoms on the Generalized Anxiety Disorder Questionnaire (GAD-7) | 10 week study period
  The GAD-7, assessed weekly, is a 7-item questionnaire of anxiety symptoms over the past week with all items on a "0" (not at all) to "3"(nearly every day) scale. Total scores range from 0 to 21; higher scores reflect greater levels of anxiety.
Change in Adaptive Behavior Assessment System - 3 (ABAS-3) | 10 week study period
  The ABAS-3 is a measure of adaptive function that yields age-standardized scores for three domains (Conceptual, Social and Practical) and an overall Global Adaptive Composite. Each domain and the overall General Adaptive Composite result in a standard score, with a mean of 100 and a standard deviation of 15 (scores between 86 and 114 are considered "Average" on this instrument; scores under 70 are classified as "Extremely Low" relative to same aged peers). Each domain is composed of several subdomains that yield scaled scale scores (Mean=10, SD=3), with scores between 7 and 13 falling in the "Average" range.
Change in Behavioral Activation for Depression Scale | 10 week study period; 4 week post-treatment
  The BADS is a 25-item measure designed to assess how clients become activated over the course of Behavior Activation treatment. There are 25 questions, each rated on a seven point scale ranging from 0 to 6. There are four subscales:
  AC = Activation subscale [score range 0 to 42] AR = Avoidance/Rumination subscale [score range 0-48] WS = Work/School Impairment subscale [score range 0-30] SI = Social Impairment subscale [score range 0-30] Higher scores indicate a better outcome on the Activation subscale. Higher scores indicate a worse outcome on the Avoidance/Rumination subscale, Work/School Impairment subscale, and Social Impairment subscale.
Change in Idiographic target goals | 10 week study period; 4 week post-treatment
  Clients are asked to identify 3 goals they would like to accomplish. There are no scores or scales. Each goal is a statement shared by the client relevant to their own experiences. Target goals are sensitive to change in treatment contexts.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No